CLINICAL TRIAL: NCT03351387
Title: Assessment of Wound Necrosis in Lower Extremity Surgery Using SPY Intra-operative Angiography
Brief Title: Wound Necrosis in Lower Extremity Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brandon James Yuan, Principal Investigator, Mayo Clinic
Other Study IDs: 17-004049
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Extremity Lower Wounds
Keywords: amputation; necrosis; high risk lower extremity wound
MeSH Terms: conditions — Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SPY Intra-operative Angiography: The SPY Fluorescent Imaging System
  Interventions: Combination Product: SPY Intra-operative Angiography

INTERVENTIONS:
Combination Product: SPY Intra-operative Angiography — The SPY Intra-operative Angiography Fluorescent Imaging System consists of an imaging head equipped with a charged coupled device (CCD) camera, a laser light source and a distance sensor. The imaging head is attached to an articulating arm on a mobile cart containing the central processing unit, keyboard, monitor, and mouse. SPY is used in tandem with indocyanine green (ICG), a water-soluble tricarbocyanine dye. Once the camera is in place, 5 cc of diluted ICG is pushed through an IV line and is flushed immediately; simultaneously the room lights must be dimmed. Perfusion images will be recorded then the SPY system will be removed from the operating room.

SUMMARY:
Researchers are performing this study to evaluate if intraoperative angiography can be shown numerically to determine which wounds are at high risk of wound necrosis/breakdown.

DETAILED DESCRIPTION:
At the beginning of the Participants surgical procedure, a picture will be obtained using intraoperative angiography using ICG dye which the camera can detect. This dye will be provided through intravenous access. The picture will be taken of the wound to determine preoperative blood flow to the area where the incision is planned. After the wound has been closed postoperatively, a final picture, using the procedure described above, will be taken to determine blood flow after closure of the wound. These images will be obtained using intraoperative angiography. The Participant will be followed after the surgical procedure at standard intervals as determined by the surgeon until the wound heals or requires further intervention.

ELIGIBILITY:
Inclusion Criteria:

-Surgical indication for high risk lower extremity surgery

Exclusion Criteria:

* Previous high risk lower extremity surgery
* Revision high risk lower extremity surgery
* Traumatic amputation
* Active infection of any kind or chronic infection with HIV, Hepatitis C, or Syphilis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: high risk lower extremity surgical candidates
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Wound necrosis | 4 weeks after surgical intervention
  Superficial wound necrosis, as evidenced by photography

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Yuan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials